CLINICAL TRIAL: NCT03102528
Title: Acute Kidney Injury After Cardiac Surgery - A Retrospective Single-center Study
Brief Title: Acute Kidney Injury Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Phyisician, University of Giessen
Other Study IDs: 79/16 D
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: All adult patients undergoing cardiac surgery (elective/emergent) at San Bortolo Hospital, Vicenza, Italy during November 2014 - October 2015
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Acute kidney injury (AKI) occurs in approximately one-third of patients undergoing cardiac surgery (CS), and represents one of the most significant negative predictors of patient outcome in this population. The investigators sought to examine the risk factors associated with the development of AKI and renal recovery in patients undergoing cardiac surgery at San Bortolo Hospital, Italy 2014-2015.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in approximately one-third of patients undergoing cardiac surgery (CS), and represents one of the most significant negative predictors of patient outcome in this population. The investigators sought to examine the risk factors associated with the development of AKI and renal recoveryin patients undergoing cardiac surgery at San Bortolo Hospital, Italy during November 2014 - October 2015.

ELIGIBILITY:
Inclusion Criteria:

- Adult cardiac surgery

Exclusion Criteria:

1. Missing baseline serum creatinine (defined as a serum creatinine value within 90 prior to surgery) or missing serum creatinine within 3 days before hospital discharge
2. Stage 5 chronic kidney disease (estimated glomerular filtration rate <15 ml/min/1.73 m2 or receipt of chronic dialysis)
3. Solid organ transplant recipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery (elective, urgent and emergent; coronary artery bypass, valve replacements, combined or other surgery, with cardiopulmonary bypass) between November 2014 and October 2015 at the Division of Cardiac Surgery, San Bortolo Hospital, in Vicenza, Italy
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute kidney injury using full Kidney Disease Improving Global Outcomes criteria | within 7 days
  Development of AKI within 7 days.

SECONDARY OUTCOMES:
Renal recovery | Within 1 month
  Defined as the absence of any stage of AKI by either serum creatinine or urine output criteria at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — International Renal Research Institute of Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryden L, Sartipy U, Evans M, Holzmann MJ. Acute kidney injury after coronary artery bypass grafting and long-term risk of end-stage renal disease. Circulation. 2014 Dec 2;130(23):2005-11. doi: 10.1161/CIRCULATIONAHA.114.010622. Epub 2014 Sep 19. PMID 25239439
- [Background] Pickering JW, James MT, Palmer SC. Acute kidney injury and prognosis after cardiopulmonary bypass: a meta-analysis of cohort studies. Am J Kidney Dis. 2015 Feb;65(2):283-93. doi: 10.1053/j.ajkd.2014.09.008. Epub 2014 Nov 5. PMID 25445101